CLINICAL TRIAL: NCT07238218
Title: Exploring the Effectiveness of Incorporated Versus Additional Dual-Task Training Program in Community Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ching-yi Wu (Other)
Collaborators: National Cheng Kung University Governance Framework for Human Research Ethics (Unknown)
Responsible Party: Sponsor-Investigator, Ching-yi Wu, Distinguished Professor and Associate Dean of College of Medicine, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 109-036
Record Dates: First submitted 2025-09-09; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Incorporated Dual-task Training; Additional Dual-task Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The motor training component (Experimental): The motor training component included stretching, aerobic exercise, strength training, and balance exercises. Exercise intensity was gradually increased to a moderate level (50-70% of participants' maximum heart rate) using low-impact modalities to minimize injury risk and was adjusted according to individual physical condition throughout the intervention. Warm-up and cool-down periods involved whole-body muscle stretching. Aerobic exercises consisted of walking, marching in place, high knee lifts, kicking motions, leg curls, touchdown steps, and box steps, combining upper and lower limb movements to produce rhythmic and repetitive patterns. Strength training comprised squats, lunges, chair sit-to-stands, weightlifting using water-filled bottles, farmer's walks, and elastic band exercises targeting both upper and lower limbs. Balance exercises included single-leg stands, heel-to-toe walking, ball kicking, and cross-stepping.
  Interventions: Behavioral: the additional dual-task training group (ADT); Behavioral: the incorporated dual-task training group (IDT)
- The cognitive training (Experimental): The cognitive training targeted domains such as attention, language, memory, calculation, and processing speed. Each session incorporated one or more cognitive domains. Attention tasks involved responding to visual or auditory cues, spotting differences in quantity, size, color, direction, or shape, and identifying specific objects within cluttered environments. Language tasks included naming fruits, animals, and vegetables, playing word solitaire, engaging in word association, constructing sentences, spelling, reading, and picture-based storytelling. Calculation tasks required solving arithmetic problems or calculating shopping list costs. Processing speed activities involved timely responses to questions, such as number comparisons. Memory tasks focused on recalling numbers, symbols, words, or daily items after presentation, as well as remembering spatial locations, shopping lists, or informational content from brochures and images.
  Interventions: Behavioral: the additional dual-task training group (ADT); Behavioral: the incorporated dual-task training group (IDT)

INTERVENTIONS:
Behavioral: the additional dual-task training group (ADT) — the cognitive task was performed concurrently but independently from the motor task, functioning as a distractor rather than a necessary prerequisite for task completion. Examples included performing lower limb strength exercises while solving arithmetic problems or reciting memorized items while stepping.
Behavioral: the incorporated dual-task training group (IDT) — the cognitive task was integrated within the motor task and was essential for successful completion of the combined motor-cognitive activity. Examples included memorizing and executing movement sequences akin to dancing or completing ladder stepping patterns in a predetermined order.

SUMMARY:
This study compared the effects of IDT and ADT on cognitive function, physical performance, instrumental activities of daily living (IADL), and quality of life in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Able to follow instructions (Mini-Mental State Examination score ≥ 20)
* Montreal Cognitive Assessment (MoCA) score > 20
* No difficulty performing basic activities of daily living
* No diagnosis of dementia confirmed by a neurologist

Exclusion Criteria:

* Self-reported diagnosis of neurological disorders
* Unstable medical conditions (e.g., recent myocardial infarction, heart failure, recent heart surgery, or severe asthma)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 164 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. Minimum: 0 (worst performance) Maximum: 30 (best performance) The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Word List (WL) subtest from the Chinese version of the Wechsler Memory Scale-Third Edition (WMS-III) | Before the intervention arms within a week, within a week after the waiting period ends, and within a week after the last treatment .
  The Word List (WL) subtest from the Chinese version of the Wechsler Memory Scale-Third Edition (WMS-III) is a standardized and reliable measure of working memory . This study utilized WL Part I (WL-I), where participants are verbally presented with a list of 12 unrelated words over four trials and asked to recall the words immediately after each trial. Raw scores represent the total number of correct recalls across trials and are converted into age-adjusted scaled scores. Higher scores reflect better memory performance. The WL-WMS has demonstrated strong internal consistency (Cronbach's alpha > 0.80) and high construct validity across diverse populations .
Change scores of Stroop Color and Word Test (SCWT) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Stroop Color and Word Test (SCWT) was used to examine inhibitory control . The primary measure used was the time difference (in seconds) between the congruent and incongruent conditions. Smaller differences indicate better inhibitory control. The Stroop test has shown high test-retest reliability (ranging between 0.70 and 0.91) and convergent validity with other executive function measures .
Change scores of Digit Symbol Substitution Test (DSST) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Digit Symbol Substitution Test (DSST), a subtest of Wechsler Adult Intelligence Scale(WAIS), was used to assess information processing speed. It is sensitive to detect cognitive impairment and changes in cognitive function . Participants are required to match symbols to corresponding numbers and copy the symbols into designated spaces within 120 seconds. The DSST score is the total number of correct symbols, with higher scores indicating better information processing speed. The DSST demonstrates excellent test-retest reliability (r = 0.89) and good concurrent validity with other cognitive processing measures .
Change scores of Timed Up and Go (TUG) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The TUG is a widely used screening tool to assess mobility and balance in community-dwelling older adults and to identify individuals at risk of falling ). Faster completion times indicate better functional mobility. The TUG demonstrates excellent inter-rater and test-retest reliability (ICC > 0.90) and good predictive validity regarding fall risk .
Change scores of Community Integration Questionnaire (CIQ) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Community Integration Questionnaire (CIQ) assesses individuals' integration into social networks and engagement in productive activities such as employment, education, or volunteer work . Higher scores indicate great level of social integration. It has shown good internal consistency (Cronbach's alpha approximately 0.70-0.80) and acceptable construct validity .
Change scores of Lawton Instrumental Activities of Daily Living(L-IADL) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Lawton IADL Scale is a valid tool designed to evaluate the ability to perform tasks and detect early functional decline. It is a reliable and valid tool commonly used for evaluating older adults with cognitive impairment . The scale measures tasks such as using a telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and financial management. Higher scores indicate greater independence in IADLs.
Change scores of Box and Block Test (BBT) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Box and Block Test (BBT) assesses gross manual dexterity . Participants move wooden blocks from one box compartment to another within 60 seconds. The number of blocks that are moved from one compartment to another compartment is recorded. The more blocks means the better gross manual dexterity. The BBT shows excellent test-retest reliability (ICC = 0.95) and strong validity for manual dexterity evaluation in older adults and clinical populations .
Change scores of Serial Sevens Test (SST) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The Serial Sevens Test (SST) evaluates working memory via serial subtraction by sevens . Correct and incorrect responses to SST are recorded, and the corrected number which is the difference between correct and incorrect responses is calculated. The more corrected numbers means the better working memory. While specific reliability data is limited, SST performance correlates moderately to strongly with other working memory and attention tasks, suggesting acceptable construct validity .
Change scores of Frequency Discrimination (FD) | Baseline, posttest(after completing the intervention,often baseline after 4 week) , Midterm(2 week after completing intervention) , 3 -month after completing intervention
  The frequency discrimination (FD) assesses sustained attention by requiring participants to distinguish between high and low auditory pitches. Participants discriminated between high (1000 Hz) and low (500 Hz) pitches and reported their answers in 18 trials conducted in 60 seconds. There was a total of 18 trials conducted in 60 s. Specifically, there were nine trials each for high- and low-pitch sounds, presented in random order with intervals of 1 to 4 seconds. Correct and incorrect responses to FD are recorded, and the corrected number which is the difference between correct and incorrect responses is calculated. Higher scores indicate better sustained attention. The task shows acceptable test-retest reliability and construct validity within auditory attention paradigms .

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan, Guishan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No